CLINICAL TRIAL: NCT03408548
Title: Effects of Probiotic Therapy in the Treatment of Periodontitis: a Study of Clinical, Microbiological and Immunological Profile of the Host Response.
Brief Title: Effects of Probiotic Therapy in the Treatment of Periodontitis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Michel Reis Messora, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 06278012.1.0000.5419
Record Dates: First submitted 2018-01-11; First posted 2018-01-24 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Periodontitis; Probiotics
Keywords: Bifidobacterium animalis subsp. lactis; Probiotic; Periodontitis treatment; Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: According to a random numeric table generated by a computer software, the study coordinator will allocate each patient into one of the following groups: Control (Scaling and Root Planing - SRP) or Test (SRP + probiotic therapy). The subjects (Control group) will receive placebo lozenge. In the Test group, the lozenge will contain Bifidobacterium lactis HN019. Individuals will be instructed (immediately after the first session of mechanical instrumentation) to consume twice a day for 4 weeks by dissolving the lozenge before bedtime and when wake up. They will also be instructed not to consume other probiotic product during the study. Clinical, immunological and microbiological parameters will be assessed at baseline (pre-intervention) and after completion of non-surgical periodontal therapy 30 and 90 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Periodontal clinical examination (pre- and post-intervention) will be conducted by a single trained and calibrated examiner, who will be blinded to the experimental groups of the study. The examiner will also be blinded to the microbiological and immunological evaluations. SRP procedures will be performed by specialist in Periodontics, trained for these purposes, who will also be blinded to the experimental groups of the study.
  The coded lozenge will be given to the examiner, who will distribute them to the patients and will not have any access to information regarding the content of the lozenge. In addition, the patients will be blinded to the content of the lozenge and the treatment assignment during the study. The meaning of each code number will be revealed by the study coordinator only after conducting the statistical analysis of the experimental data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Scaling root planning + two lozenge per day not containing Bifidobacterium animalis lactis HN019 for 30 days.
  Interventions: Procedure: Scaling root planning; Other: Placebo
- Probiotic (Experimental): Scaling root planning + two lozenge per day containing Bifidobacterium animalis lactis HN019 (10x9 colony-forming units) for 30 days.
  Interventions: Procedure: Scaling root planning; Dietary Supplement: Probiotic

INTERVENTIONS:
Procedure: Scaling root planning — Periodontal treatment
Dietary Supplement: Probiotic — two lozenge per day containing Bifidobacterium animalis lactis HN019
  Arms: Probiotic
Other: Placebo — two lozenge per day not containing Bifidobacterium animalis lactis HN019
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the effect of the probiotic therapy as an adjunct to non-surgical periodontal treatment in patients diagnosed with Generalized Chronic Periodontitis. Clinical study's hypothesis is that with the use of probiotic therapy, the standard treatment could be enhance.

DETAILED DESCRIPTION:
Before the study begins, the selected individuals will be identified by a numeric code and will receive instructions regarding oral hygiene as well as supragingival scaling in all teeth. According to a random numeric table generated by a computer software, the study coordinator will allocate each patient into one of the following groups: Control (Scaling and Root Planing - SRP) or Test (SRP + probiotic therapy). The subjects (Test and Control groups) will receive lozenge containing/not containing. In the Test group, the lozenge will present Bifidobacterium lactis HN019 (HN019). Individuals will be instructed (immediately after the first session of mechanical instrumentation) to consume twice a day for 4 weeks by dissolving the lozenge before bedtime, and when wake up. They will also be instructed not to consume other probiotic product during the study. Clinical, immunological and microbiological parameters will be assessed at baseline (pre-intervention) and after completion of non-surgical periodontal therapy 30 and 90 days. All patients will receive detailed information regarding the study (goals, benefits and risks) according to the Term of Consent. The sample size was determined using the software Graphpad Statemate 2.0 (GraphPad Software, Inc., San Diego, CA, USA). The ideal sample size to ensure an 80% power in the statistical analysis of the data obtained in this study was calculated considering the differences of means and standard deviations between the test and control groups of the study by Vivekananda et al. (2010). The α value was set at 0.05. The average dropout of patients in our previous studies (approximately 20%) was also considered to calculate the sample size. Thus, a sample size of at least 30 patients was considered appropriate for this study. The normality and homoscedasticity of the data obtained will be checked. Comparisons within groups and among groups at different time intervals will be performed through parametric or non-parametric appropriate tests. The significance level will be set at 5% in all tests. All calculations will be performed by SPSS software (SPSS, Chicago IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* More than 30 years old
* All patients must present good general health.
* Previously untreated periodontitis
* Minimum of 15 teeth

Exclusion Criteria:

* Having received antibiotics for any purpose within 6 months prior to entering the study or the need for antibiotic coverage for dental treatment
* Pregnancy and nursing
* Acute oral lesions or necrotizing ulcerative periodontitis,
* A history of diabetes, rheumatic fever, liver or kidney disease, neurological deﬁciencies, immunological diseases or use of medication which may affect periodontal tissue, (phenytoin, cyclosporin, niﬁdepine, chronic use of non-steroidal anti-inﬂammatory drugs)
* Current smoker or former smoker

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
Changes in probing depth. | Baseline, 30 days, 90 days.
  millimeter.

SECONDARY OUTCOMES:
Changes in plaque index. | Baseline, 30 days, 90 days.
  sites.
Changes in the levels of interleukin(IL)-1βeta, IL-8 and IL-10 in the gingival crevicular fluid. | Baseline, 30 days, 90 days.
  pg/ml.
Changes in the levels of immunoglobulin A in saliva. | Baseline, 30 days, 90 days.
  mg/dL.
Changes in the subgingival microbiota. | Baseline, 30 days, 90 days.
  mean count.
Changes in the expression of beta-defensin-3, toll like receptor-4, cluster of differentiation (CD)-4 and CD-8. | Baseline, 30 days.
  cells/mm2
Changes in the attachment level. | Baseline, 30 days, 90 days.
  millimeter.
Changes in bleeding on probing. | Baseline, 30 days, 90 days.
  sites.

CONTACTS AND LOCATIONS:
Overall Officials: Michel R Messora, Phd, Principal Investigator — University of Sao Paulo - FORP
Locations (1):
- School of Dentistry of Ribeirão Preto - University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laleman I, Yilmaz E, Ozcelik O, Haytac C, Pauwels M, Herrero ER, Slomka V, Quirynen M, Alkaya B, Teughels W. The effect of a streptococci containing probiotic in periodontal therapy: a randomized controlled trial. J Clin Periodontol. 2015 Nov;42(11):1032-41. doi: 10.1111/jcpe.12464. Epub 2015 Nov 29. PMID 26427036
- [Background] Matsubara VH, Bandara HM, Ishikawa KH, Mayer MP, Samaranayake LP. The role of probiotic bacteria in managing periodontal disease: a systematic review. Expert Rev Anti Infect Ther. 2016 Jul;14(7):643-55. doi: 10.1080/14787210.2016.1194198. Epub 2016 Jun 3. PMID 27224284
- [Background] Messora MR, Oliveira LF, Foureaux RC, Taba M Jr, Zangeronimo MG, Furlaneto FA, Pereira LJ. Probiotic therapy reduces periodontal tissue destruction and improves the intestinal morphology in rats with ligature-induced periodontitis. J Periodontol. 2013 Dec;84(12):1818-26. doi: 10.1902/jop.2013.120644. Epub 2013 Jan 17. PMID 23327675
- [Derived] Invernici MM, Furlaneto FAC, Salvador SL, Ouwehand AC, Salminen S, Mantziari A, Vinderola G, Ervolino E, Santana SI, Silva PHF, Messora MR. Bifidobacterium animalis subsp lactis HN019 presents antimicrobial potential against periodontopathogens and modulates the immunological response of oral mucosa in periodontitis patients. PLoS One. 2020 Sep 22;15(9):e0238425. doi: 10.1371/journal.pone.0238425. eCollection 2020. PMID 32960889
- [Derived] Invernici MM, Salvador SL, Silva PHF, Soares MSM, Casarin R, Palioto DB, Souza SLS, Taba M Jr, Novaes AB Jr, Furlaneto FAC, Messora MR. Effects of Bifidobacterium probiotic on the treatment of chronic periodontitis: A randomized clinical trial. J Clin Periodontol. 2018 Oct;45(10):1198-1210. doi: 10.1111/jcpe.12995. Epub 2018 Sep 24. PMID 30076613